CLINICAL TRIAL: NCT05134870
Title: Mimic-game & Groove: A TeleXercise Intervention to Get Active & Get Healthy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Tanvi Bhatt, PI, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0923
Record Dates: First submitted 2021-08-13; First posted 2021-11-26 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Healthy Older Adults
Keywords: Tele-rehabilitation; TeleXercise; Mimic-Game-&Groove
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TeleXercise intervention (Experimental): TeleXercise intervention will be delivered via exergaming-based animation videos combined with or without cognitive exercises by a health coach. Participants will need a computer/tablet/smart phone for the study. The health coach will launch the exercise application on their computer and share their screen with the participants. They have to mimic the exercises shown to them. The intervention will have 12 sessions for 4 weeks, each session for 1.5 hours, including warm-ups and cool-down. Warm-up and cool down are for 20 minutes. A wearable device provided will measure the heart rate and physical activity during the training. Participants are provided with a set of balance exercises which includes non-interactive balance games (stepping forward, backward, sideways), Tai-Chi, Weight shifting (to right leg, left leg and practice distributing equal weights on both the legs), Aerobic (stepping in place), dance, strength, and stretching
  Interventions: Behavioral: Mimic- game and groove- Telerehabilitation

INTERVENTIONS:
Behavioral: Mimic- game and groove- Telerehabilitation — Participants will mimic the exergaming-based animation videos shown to them by the health coach. They will also wear a wearable device that will measure the heart rate and physical activity during the training. The intervention will have 12 sessions for 4 weeks, each session for 1.5 hours, including warm-ups and cool-down. Warm-up and cool down are for 20 minutes. Additionally, Participants are provided with a set of balance exercises which includes non-interactive balance games (stepping forward, backward, sideways), Tai-Chi, Weight shifting (to right leg, left leg and practice distributing equal weights on both the legs), Aerobic (stepping in place), dance, strength, and stretching
  Other Names: Tele rehabilitation

SUMMARY:
The composite effect of reduced balance, cognition, gait abnormalities/gait disturbances, and physical activity in older adults leads to fear of falling and decreased participation in daily activities, resulting in reduced cardiovascular fitness and deconditioning. Although many conventional balance and strength training programs have been implemented for older adults, these adults do not receive adequate practice dosage to make significant improvements, most likely due to lack of adherence to therapy and/or inadequate incorporation of all domains of the ICF model (body functions and structures, activities and participation) and lack of targeting cognitive-motor interference (deterioration of motor and/or cognitive function when both tasks are performed together). The use of TeleXercise via Tele rehabilitation has been found to be relatively enjoyable for older adults due to increased motivation and adherence to therapy, which led to the added improvement of physical and cognitive functioning. The overall aim of this pilot is to develop and test the Mimic-Me & Groove TeleXercise platform and then evaluate the compliance and efficacy of the TeleXercise intervention compared to control group receiving standard of care (education on conventional exercise and fall prevention program) for older adults as well as its effect on enhancing balance, gait, and cognition, and physical activity. Investigators also hope that the net effect of improvement in these domains of health outcomes will result in pre and post improvement in endurance and cardiovascular function and reduction of fall risk and improved quality of life of older adults. The study investigates the efficacy of a TeleXercise intervention in older adults by demonstrating its feasibility, compliance rate and also determine the efficacy of the Mimic-Me & Groove TeleXercise in improving health outcomes such as motor and cognitive functions, thereby reducing cognitive-motor interference. The study will also aim to determine the effectiveness of the TeleXercise in improving cardiovascular fitness and physical activity (PA) in older adults.

DETAILED DESCRIPTION:
Aging results in neuromuscular deterioration, such as impaired balance control, gait instability, and worsening cognition with increasing evidence pointing to the over-reliance on cognitive function to perform even simple motor tasks. Such deterioration has been shown to affect daily functional activities, quality of life, and cardiovascular fitness, along with an increase in the risk of falling. Physical activity has been recommended as a means to slow down neuromuscular deterioration and enhance gait, stability, and cognition in older adults. Further, increased levels of physical activity have also demonstrated positive effects on cardiovascular fitness (heart rate variability, HRV).However, older adults do not meet the recommended daily requirement (of at least 5000 steps/day) due to reduced motivation and lack of compliance to physical activity regimen. The lack of compliance may emanate from difficulty to commute to outpatient rehabilitation centers, lack of involvement, and the decreased participatory nature of most conventional physical therapy interventions. As a result, there is the need to implement a home-based TeleXercise intervention for older adults. This TeleXercise intervention should be motivational and enjoyable with increased participation or involvement, while aiming to improve cognition, physical activity and balance for fall prevention in older adults. Exercise training provided via Tele rehabilitation, as an alternative therapy, has shown to increase balance control and gait as well as increase motivation among older adults. Further, our preliminary studies conducted in the laboratory has shown promising results on various alternative methods for rehabilitating older adults. Among which exergaming-based dance therapy has exhibited feasibility in improving balance, mobility and cardiovascular function, along with decreasing fall risk. Also, older adults exhibit deterioration of balance control and gait in dual-task conditions (i.e., simultaneous performance of two tasks). Few systematic reviews have emphasized on some task-specific exercises to improve balance control in older adults, such as single leg stance, modified tree pose etc. Thus, it could be postulated that older adults could benefit from an integrated comprehensive therapy program which incorporates various physical exercises, such as conventional methods of balance exercises, exergaming-based balance games, and dance with cognitive training. However, there is no data on the feasibility and effect of such comprehensive therapy on efficacy, compliance, balance, cognitive, gait and physical activity measures among older adults. Given that older adults lack compliance to therapy, investigators therefore, seek to examine the feasibility of a comprehensive TeleXercise-based intervention through the use of a comprehensive intervention protocol incorporating various physical exercises. Specifically, task-specific balance training provided via observing and imitating an exercise activates Action Observation Network system (AON) and other brain centers, which is known to improve balance control through increased plasticity of neural systems (mirror neurons) for optimal observation and actual performance of movement.

Aim1: The study will test the applicability, feasibility and compliance of TeleXercise intervention (N=17) to improve physical function and reduce fall-risk in community-dwelling older adults.

Hypothesis: Participants will tolerate the training paradigm and will demonstrate significant improvements in balance, gait, cardiovascular and cognitive performance under single and dual-task conditions. Participants will also demonstrate appropriate compliance (attend >24/30 session) and motivation (>Intrinsic Motivation Inventory scores) post-intervention.

Aim 2: To examine if the proposed TeleXercise intervention will lead to higher cognitive function post-intervention.

Hypothesis: Participants will show significantly greater global cognitive function, executive and working memory and decreased cognitive-motor load post-training compared to pre-training

Aim 3: To determine the effect of TeleXercise intervention on improving physical fitness (physical activity, PA) of community-based older adults.

Hypothesis 3: Post-training measures will depict a significant improvement in physical activity fitness.

Ancillary hypothesis: To determine if improved cognitive-motor function and physical fitness gained from a TeleXercise intervention will translate into improved falls efficacy, quality of life and physical activity post withdrawal of intervention with reduced fatigue and exertion.

Hypothesis: At 8 weeks (4 weeks post-intervention or withdrawal), participants will have retention of the post-training gains in single and dual-task conditions and cardiovascular fitness, which will translate into improved falls efficacy (improvement on Activities-specific Balance Confidence scale), quality of life (Older People's Quality of Life Questionnaire (OPQOL-35) and participation (improved Community Integration Scale) compared to their pre-training. Participants will also show improved falls efficacy translated to improved community ambulation (physical activity) and reduced fatigue and exertion (Borg Scale, NASA TLX scale)

ELIGIBILITY:
Inclusion Criteria:

1. Age group: Community-dwelling healthy older adults between the age group of 55 - 85 years
2. Participants without any history of fracture for the last 1 year
3. Should have either a desktop computer/laptop/tablet and a WIFI connection.
4. Absence of any acute or chronic neurological (Stroke, Parkinson's disease, Alzheimer's disease), cardiopulmonary, musculoskeletal, or systemic diagnosis.
5. No recent major surgery (< 6 months) or hospitalization (< 3 months)
6. Not on any sedative drugs
7. Can understand and communicate in English

Exclusion Criteria:

1. Participants will not proceed with the study if at baseline measurement HR > 85% of age-predicted maximal heart rate (HRmax) (HRmax = 220 - age)
2. Inability to stand for at least 5 minutes without an assistive device (length of each exercise)
3. History of bone fracture or significant other systemic disease or surgery in the last six months
4. Uncontrolled acute medical, surgical, neurological or cardiovascular disease.
5. Moderate to severe cognitive impairment (MOCA <24/30)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Change in time during 30-second chair stand test. | Change in time from pre-test (Week 0) to post-training (week 5)
  This test is conducted to assess leg strength and endurance.
Change in time during four-step square test | Change in time from pre-test (Week 0) to post-training (week 5)
  To test the dynamic balance and to assess the person's ability to step over objects forward, sideways, and backwards
Change in time during Sharpened Romberg | Change in time from pre-test (Week 0) to post-training (week 5)
  To assess the static balance of participants in sensory integration taxing condition
Change in time during 2-minute step in place test | Change in time from pre-test (Week 0) to post-training (week 5)
  To assess the cardiovascular exercise tolerance
Change in time during One-legged Stance test | Change in time from pre-test (Week 0) to post-training (week 5)
  To assess the static balance of participants in sensory integration taxing condition
Change in time during Tinetti Performance Oriented Mobility Assessment | Change in time from pre-test (Week 0) to post-training (week 5)
  To assess gait and balance together

SECONDARY OUTCOMES:
Change in correct responses during Letter Number sequencing test | Change in number of correct response from pre-test (Week 0) to post-training (week 5)
  To assess cognitive performance
Change in correct responses during Visual stroop test | Change in number of correct response from pre-test (Week 0) to post-training (week 5)
  To assess cognitive performance
Change in correct responses during Auditory stroop | Change in number of correct response from pre-test (Week 0) to post-training (week 5)
  To assess cognitive performance
Change in correct response during Flanker inhibitory control and attention test | Change in number of correct response from pre-test (Week 0) to post-training (week 5)
  To assess cognitive performance
Change in correct response during List Sorting Memory test | Change in number of correct response from pre-test (Week 0) to post-training (week 5)
  To assess cognitive performance
Change in correct response during Dimensional Change card sort test | Change in number of correct response from pre-test (Week 0) to post-training (week 5)
  To assess cognitive performance
Change in correct response during Pattern comparison Processing speed test | Change in number of correct response from pre-test (Week 0) to post-training (week 5)
  Evaluates the processing speed of cognitive functioning.
Change in score of Physical Activity Scale for elderly | Change in score from pre-test (Week 0) to post-training (week 5)
  To assess self-reported measure of physical activity
Change in score of Activities Specific Balance Confidence scale (ABC scale) | Change in score from pre-test (Week 0) to post-training (week 5)
  To assess self-reported measure of balance confidence. Scores range from 0-100. Score of zero represents no confidence, a score of 100 represents complete confidence.
Change in score of Older People's Quality of Life Questionnaire (OPQOL-35) | Change in score from pre-test (Week 0) to post-training (week 5)
  To assess their quality of life. There are 35 items, with scores ranging from 35- 175. Lesser scores indicate better quality of life, while higher scores indicate reduced quality of life.
Change in score of Community Integration Scale (CIS). | Change in score from pre-test (Week 0) to post-training (week 5)
  To assess their participation in the community. Total score range from 0-29. High scores indicate greater independence and social integration
Change in score of Modified Borg Scale (MB) | Change in score from pre-test (Week 0) to post-training (week 5)
  To determine the exertion and fatigue level during the training session and during pre-and post-assessment. Scores range from 0-10. Scale rates the difficulty breathing. It starts at number 0 where breathing is causing no difficulty at all and progresses through to number 10 where breathing difficulty is maximal.
Change in score of NASA Task Load Index scale (NASA-TLX) | Change in score from pre-test (Week 0) to post-training (week 5)
  To determine the physical and cognitive load during the training session as well during pre- and post-assessment. The score ranges from1-20, where lowers scores indicate less demand, and higher scores indicate increased demand.

CONTACTS AND LOCATIONS:
Overall Officials: Tanvi S Bhatt, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States